CLINICAL TRIAL: NCT05007613
Title: A Single-arm Phase II Study of Cabozantinib and Atezolizumab in Patients With Recurrent or Metastatic Esophageal Squamous Cell Carcinoma Who Failed a Platinum-based Chemotherapy
Brief Title: Second-line Cabozantinib and Atezolizumab in Patients With Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ipsen (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202101041MIPB
Record Dates: First submitted 2021-07-14; First posted 2021-08-16 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Cancer; Metastatic Cancer; Squamous Cell Carcinoma
Keywords: esophageal cancer; squamous cell carcinoma; cabozantinib; atezolizumab; immune checkpoint inhibitor
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasm Metastasis; Carcinoma, Squamous Cell | interventions — cabozantinib; atezolizumab

STUDY DESIGN:
Intervention Model Description: cabozantinib and atezolizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- cabozantinib plus atezolizumab (Experimental): cabozantinib 40mg PO QD atezolizumab 1200mg IVD 30-60mins Q3W
  Interventions: Drug: Cabozantinib 40 MG; Drug: Atezolizumab Injection

INTERVENTIONS:
Drug: Cabozantinib 40 MG — Cabozantinib (Cabometyx) 40 MG PO QD
  Other Names: Cabometyx
Drug: Atezolizumab Injection — atezolizumab (Tecentriq) 1200mg IVF 30-60mins Q3W
  Other Names: Tecentriq

SUMMARY:
To demonstrate that combination of cabozantinib and atezolizumab is safe and efficacious in patients with recurrent/metastatic esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Patients with histologically proven squamous cell carcinoma of esophagus and had progression from first-line platinum-based chemotherapy for recurrent or metastatic ESCC, or progression within 6 months after neoadjuvant, definitive, or adjuvant chemo(radio) -therapy for loco-regional ESCC would be eligible for this trial. Eligible patients will receive daily 40mg cabozantinib plus i.v. atezolizumab 1200mg Q3W for treatment response evaluation. Primary endpoint is the objective response rate, and secondary endpoints include progression-free survival, overall survival, and safety profiles.

ELIGIBILITY:
Inclusion Criteria:

* 1.Histologically proven squamous cell carcinoma of esophagus.
* 2.Progression from first-line platinum-based chemotherapy for recurrent or metastatic ESCC, or progression within 6 months after neoadjuvant, definitive, or adjuvant chemo(radio) -therapy for loco-regional ESCC.
* 3.Measurable disease per RECIST 1.1
* 4.Recovery to baseline or ≤ Grade 1 per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy as determined by the Investigator.
* 5.Age twenty years or older
* 6.Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* 7.The subject is receiving antiviral therapy per local standard of care if the subject has active HBV infection (defined by HBsAg positive); the subject must have HBV DNA < 500 IU/mL.Patients with HBV infection are required to continue antiviral therapy throughout the Treatment Period, and till at least 3 months after discontinuing Trial treatment.
* 8.Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days prior to treatment:
* Absolute neutrophil count (ANC) ≥ 1500/µL without granulocyte colony-stimulating factor support within 2 weeks before screening laboratory sample collection.
* White blood cell (WBC) count ≥ 2500/µL.
* Platelets ≥ 100,000/µL without transfusion within 2 weeks before screening laboratory sample collection.
* Hemoglobin ≥ 9 g/dL without transfusion within 2 weeks before screening laboratory sample collection.
* Alanine aminotransferase (ALT), AST, and alkaline phosphatase (ALP) ≤ 3 × upper limit of normal (ULN).
* Total bilirubin ≤ 1.5 mg/dL.
* Serum albumin ≥ 2.8 g/dL.
* Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance ≥ 40 mL/min (≥ 0.67 mL/sec) using the Cockcroft-Gault equation:

Males: (140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72) Females: [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85

* Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol), or 24-h protein ≤ 1 g.
* 9.Capable of understanding and complying with the protocol requirements and must have signed the informed consent document prior to any screening assessment except those procedures performed as standard of care within the screening window.
* 10.Sexually active fertile subjects and their partners must agree to use highly effective methods of contraception that alone or in combination result in a failure rate of less than 1% per year when used consistently and correctly (see Appendix G) during the course of the study and for 5 months after the last dose of study treatment. An additional contraceptive method, such as a barrier method (eg, condom), is recommended.
* 11.Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.

Exclusion Criteria:

* 1.Previously treated with PD-1/PD-L1 blockade or any type of small molecule kinase inhibitor (including investigational kinase inhibitor)
* 2.Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
* 3.Prior radiotherapy regimen exceeding 70 Gy for a single site, including ESCC or other metastatic sites:
* For radiotherapy to treat ESCC:

If the radiation is combined with chemotherapy, a minimum of 4 months must elapse between the end of radiotherapy and registration. If the radiation is given alone, a minimum of 8 weeks must elapse between the end of radiotherapy and registration.

* For radiotherapy to treat metastatic site:

A minimum of 3 weeks must elapse between prior radiation and registration.

* All treatment areas should be fully healed with no sequelae from RT that would predispose to fistula formation. Unhealed or with sequelae from RT that would predispose to fistula formation.
* 4.Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.
* 5.Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel), except for the following allowed anticoagulants:

  1. Low-dose aspirin for cardioprotection (per local applicable guidelines) is permitted.
  2. Low-dose low molecular weight heparins (LMWH) are permitted.
  3. Anticoagulation with therapeutic doses of LMWH is allowed in subjects without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* 6.Administration of a live, attenuated vaccine within 30 days prior to treatment.
* 7.Any subject who cannot be evaluated by computed tomography (CT) because of allergy or other contraindication to both CT and MRI contrast agents.
* 8.The subject has uncontrolled, significant intercurrent or recent (within the last 3 months before treatment [unless otherwise specified below]) illness including, but not limited to, the following conditions:
* Cardiovascular disorders:

  a.Congestive heart failure (CHF) class III or IV as defined by the New York Heart Association, unstable angina pectoris, serious cardiac arrhythmias.

  b.Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.

  c.Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event or thromboembolic event (eg, DVT, pulmonary embolism) within 6 months before treatment.
* Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

  1. Tumors invading the GI-tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction.
  2. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months prior to treatment. Complete healing of an intra-abdominal abscess must be confirmed prior to treatment.
  3. Any episodes of GI bleeding requiring transfusion or hospitalization for at least 6 months before treatment.
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 3 months before treatment.
* Cavitating pulmonary lesion(s) or known endobronchial invasion.
* Lesions invading major blood vessel, including, but not limited to: inferior vena cava, pulmonary artery, or aorta.
* Other clinically significant disorders such as:

  a.Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, psoriatic arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix C for a more comprehensive list of autoimmune diseases and immune deficiencies). Subjects with the following conditions are eligible for the study: i. A history of autoimmune-related hypothyroidism and on thyroid replacement hormone ii. Controlled Type 1 diabetes mellitus and on an insulin regimen iii. Asthma that requires intermittent use of bronchodilators iv. Eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only provided all of following are true:
* Rash covers < 10% of body surface area
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months b. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days before treatment.

Note: Inhaled, intranasal, intra-articular, and topical corticosteroids and mineralocorticoids are permitted.

Transient use of systemic corticosteroids for allergic conditions such as contrast allergy is allowed.

c. Active infection requiring systemic treatment, known history of infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome d. (AIDS)-related illness, or a known positive test for tuberculosis due to tuberculosis infection. Subjects with active hepatitis B virus infection controlled with antiviral therapy are eligible (see Inclusion Criterion 7). Subjects with active, uncontrolled hepatitis C virus infection are eligible provided liver function meets eligibility criteria and are receiving management of the disease per local institutional practice (note: antiviral treatment for HCV is allowed).

e. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan f. Serious non-healing wound/ulcer/bone fracture. g.Malabsorption syndrome. h.Free thyroxine (FT4) outside the laboratory normal reference range. Asymptomatic subjects with FT4 abnormalities can be eligible.

i. Requirement for hemodialysis or peritoneal dialysis. j. History of solid organ transplant including allogeneic stem cell transplant.

* 9.Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks before treatment. Minor surgeries within 10 days before treatment. Subjects must have complete wound healing from major surgery or minor surgery before treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* 10.Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before treatment.

Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility

* 11.History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
* 12.Pregnant or breastfeeding females.
* 13.Inability to swallow tablets.
* 14.Previously identified allergy or hypersensitivity to components of the study treatment formulations or history of severe hypersensitivity to monoclonal antibodies.
* 15.Any other active malignancy at time of treatment or diagnosis of another malignancy within 2 years before treatment that requires active treatment, except for superficial skin cancer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | at least 3 weeks after the first treatment
  Overall response rate (ORR) is the proportion of patients whose tumor is significantly reduced.

SECONDARY OUTCOMES:
Progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Progression-free survival (PFS) is the time from enrollment to the first occurrence of disease progression or death from any cause (whichever occurs first) and will be conducted in the whole study population. It is designed to include progression events as determined by the investigators per RECIST 1.1 or death.
Overall survival | From date of randomization until the date of death from any cause, assessed up to 60 months
  Overall survival (OS) is the time from enrollment to death of any cause or the last follow-up (censored).
Safety (treatment-related adverse effects) | From the first treatment to 30 days after the end of study.
  The incidence and severity of toxicity will be summarized according to the NCI Common Toxicity Criteria Version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT05007613/Prot_SAP_000.pdf